CLINICAL TRIAL: NCT04209881
Title: Evaluation of Ovarian Reserve Using Anti-müllerian Hormone and Antral Follicle Count in Ankylosing Spondylitis: Preliminary Study
Brief Title: Ovarian Reserve and Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Principal investigator, Pınar kadirogullari, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019/456.14.10.2019
Record Dates: First submitted 2019-12-19; First posted 2019-12-24 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Ovarian Diseases; Ankylosing Spondylitis; Anti-Mullerian Hormone Deficiency
Keywords: Ankylosing spondylitis; fertility; anti-müllerian hormone; ovarian reserve
MeSH Terms: conditions — Ovarian Diseases; Spondylitis, Ankylosing | interventions — Ovarian Reserve; HLA-B Antigens; Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Ankylosing spondylitis: Women Who Are Diagnosed With Ankylosing Spondylitis Will Form The Study Group. Clinical And Laboratory Parameters Will Be Evaluated For Ovarian Capacity Of These Women.In order to evaluate the ovarian reserve of the patients, the parameters we routinely look at will be evaluated as follows. the results of these tests will be observed.
  Amh Will Be Looked For (Pmol / L). Antral Folukul Census In The Overin Folukular Stage Will Be Valued As Number. Fsh (Iu / L) And Estradiol (Pmol / L) Values Will Also Be Recorded.
  Interventions: Other: ovarian reserve for Ankylosing spondylitis and control groups
- Healthy women as controls: Regular menstruation with intervals of 21-35 days; cycle length variations <4 days; and both ovaries still present healthy women will create the control group.In order to evaluate the ovarian reserve of the patients, the parameters we routinely look at will be evaluated as follows. the results of these tests will be observed.
  Amh will be looked for. (pmol / l). Antral folukul census in the overin folukular stage will be valued as number. Fsh (iu / l) and Estradiol (pmol / l) values will also be recorded.
  Interventions: Other: ovarian reserve for Ankylosing spondylitis and control groups

INTERVENTIONS:
Other: ovarian reserve for Ankylosing spondylitis and control groups — Additional organ diseases due to the pathophysiology of the disease may be seen in women with ankylosing spondylitis. therefore, we established the first group of women with the diagnosis of ankylosing spondylitis.
  Women Who Are Diagnosed With Ankylosing Spondylitis Will Form The Study Group. and health women will be control group.
  Clinical And Laboratory Parameters Will Be Evaluated For Ovarian Capacity Of These Women.
  Amh Will Be Looked For (Pmol / L). Antral Folukul Census In The Overin Folukular Stage Will Be Valued As Number. Fsh (Iu / L) And Estradiol (Pmol / L) Values Will Also Be Recorded.

SUMMARY:
The aim of this study was to determine the status of ovarian reserve in patients with ankylosing spondylitis (AS) using anti-mullerian hormone (AMH) level and antral follicle count (AFC). Women with AS and women controls diagnosed according to the classification criteria proposed by the American-European Consensus Group will be included in the study. Ovarian reserve will be evaluated in terms of clinical findings, AFC and serum AMH and reproductive hormone levels.

Researchers predict that the ovarian reserve may be reduced in patients with AS due to the autoimmune process and the pathophysiology of the disease. Serum AMH and ovarian AFC may be useful for assessing ovarian reserve. It is aimed to determine the course of ovarian reserve abnormalities and the best possible biomarkers of reduced ovarian reserve in patients with AS.

ELIGIBILITY:
Inclusion Criteria:

* regular menstruation with intervals of 21-35 days;
* cycle length variations <4 days;
* both ovaries still present

Exclusion Criteria:

* history of liver failure;
* diagnosed malignancy;
* cigarette smoking;
* chronic renal failure;
* known infertility;
* presence of gynecological abnormalities such as abnormal uterine bleeding or menorrhagia;
* history of ovarian surgery;
* history of hormone preparation (including corticosteroids) use or use of herbal products within 3 months;
* diagnosis of polycystic ovary syndrome.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women who are diagnosed with ankylosing spondylitis will form the study group.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
anti-müllerian hormone (AMH) | 3 days
  For ovarian capacity AMH will be examined and AMH levels will be recorded in pmol/l
antral follicle count (AFC) | 1 day
  For ovarian capacity AFC will be examined and It will be recorded as a NUMBER.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yalcin Bahat P, Kadirogullari P, Topbas Selcuki NF, Yucel B, Cakmak K, Ureyen Ozdemir E. Ovarian reserve in patients with ankylosing spondylitis. Arch Gynecol Obstet. 2021 Jan;303(1):189-193. doi: 10.1007/s00404-020-05824-8. Epub 2020 Oct 8. PMID 33030584